CLINICAL TRIAL: NCT03738384
Title: Knee Connect: Physiotherapy Exercise Performance With Visual Feedback After Total Knee Arthroplasty - Pilot Study
Brief Title: Knee Connect: Physiotherapy Exercise Performance With Visual Feedback After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 03KINERIS2018
Record Dates: First submitted 2018-10-26; First posted 2018-11-13 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2021-03

CONDITIONS: Arthroplasty; Replacement; Knee
Keywords: Rehabilitation, Visual, Feedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TKR Patients (Experimental): Any patient 3-6 weeks post-op from a TKR
  Interventions: Device: Knee Connect + Visual Feedback System

INTERVENTIONS:
Device: Knee Connect + Visual Feedback System — A device to measure knee angle. It sends data a smartphone or tablet to be displayed as part of a visual feedback system.

SUMMARY:
The main objective of this pilot study is to determine if using a portable, accelerometer based, visual feedback system improves exercise quality. The secondary objective of this study is to investigate the effect of motivational targets by testing the effects of increasing Range of Motion (ROM) targets. The results from this study will be used to improve the visual feedback system of the Knee Connect system and serve as starting point for a larger clinical study.

DETAILED DESCRIPTION:
The research team will recruit 10 post-op total knee replacement patients who are enrolled in the Knee Class at Sunnybrook Holland Orthopaedic and Arthritic Centre to perform five exercises over two sessions. Each patient will complete five tasks.

1. Quarter squats
2. Standing hip flexion
3. Standing knee flexion
4. Sitting knee extension
5. Sitting knee flexion

The first three exercises will be performed with and without visual feedback. During standing hip flexion, standing knee flexion and quarter squat exercises, patients will first perform a set of each exercise following an instruction brochure. Patients will then repeat these exercises with the Knee Connect visual feedback system. The KneeConnect will be worn during the entire session, and will record the patient's knee angle and velocity regardless of visual feedback condition.

For the next two exercises, sitting knee extension and sitting knee flexion, patients will perform the first set of exercises (3 repetitions) with visual feedback of their leg position in space but without seeing an end target. The Knee Connect will measure the knee angle during these tests. For the subsequent set, the Knee Connect system will present a visual target for the patient to achieve. This target will be 5 degrees above the patient's maximum terminal knee angle recorded without motivational targets. A third set will be completed with the knee angle target set 10 degrees above the patient's maximum. A caveat to the target modification for seated knee extensions is that target changes to hyperextension, will result in a full extension target.

After each participant has completed the exercises with the KneeConnect system they will be asked to complete a short survey. The survey has been designed to assess the KneeConnect's usefulness and how much participants liked using the system.

After the data collection has been completed each day, the data will be transferred from the smartphone to a secure computer. These files will then be extracted to measure:

* Knee angle during each exercise
* Knee angular velocity during each exercise

A Leven's test will be used on all of the data to assess the equality of variance in each group. Each pair of data will be compared using a paired t-test to test the difference between with/without visual feedback and with/without motivational targets.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled in the "Knee Class" postoperative physiotherapy
* Be able to provide informed consent
* 3-6 weeks post-operative from primary total knee replacement surgery

Exclusion Criteria:

* Revision total knee arthroplasty
* Neuromuscular disorder
* Knee Stiffness (knee flexion of <90 degrees during previous Knee Class session)
* Hip Stiffness (hip flexion of <90 degrees)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Knee angle (degrees) | One set of measurements 3-6 weeks post TKR
  The difference in measured knee angle with and without visual feedback.
Knee velocity (degrees/s) | One set of measurements 3-6 weeks post TKR
  The difference in measured knee velocity with and without visual feedback.

SECONDARY OUTCOMES:
Peak knee flexion and extension angle (degrees) | One set of measurements 3-6 weeks post TKR
  The weekly knee range of motion (in degrees) measured by the Knee Connect

CONTACTS AND LOCATIONS:
Overall Officials: David Wasserstein, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Holland Orthopaedic & Arthritic Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Manniche C, Hesselsoe G, Bentzen L, Christensen I, Lundberg E. Clinical trial of intensive muscle training for chronic low back pain. Lancet. 1988 Dec 24-31;2(8626-8627):1473-6. doi: 10.1016/s0140-6736(88)90944-0. PMID 2904582
- [Background] Nwuga, G., & Nwuga, V. (1985). Relative therapeutic efficacy of the Williams and McKenzie protocols in back pain management. Physiotherapy practice, 1(2), 99-105.
- [Background] Kohles S, Barnes D, Gatchel RJ, Mayer TG. Improved physical performance outcomes after functional restoration treatment in patients with chronic low-back pain. Early versus recent training results. Spine (Phila Pa 1976). 1990 Dec;15(12):1321-4. doi: 10.1097/00007632-199012000-00016. PMID 2149211
- [Background] Friedrich M, Cermak T, Maderbacher P. The effect of brochure use versus therapist teaching on patients performing therapeutic exercise and on changes in impairment status. Phys Ther. 1996 Oct;76(10):1082-8. doi: 10.1093/ptj/76.10.1082. PMID 8863761
- [Background] Lam, A. W., Varona-Marin, D., Li, Y., Fergenbaum, M., & Kulić, D. (2016). Automated rehabilitation system: Movement measurement and feedback for patients and physiotherapists in the rehabilitation clinic. Human-Computer Interaction, 31(3-4), 294-334.
- [Background] Lam AW, HajYasien A, Kulic D. Improving rehabilitation exercise performance through visual guidance. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:1735-8. doi: 10.1109/EMBC.2014.6943943. PMID 25570311
- [Background] Chkeir, A., Jaber, R., Hewson, D. J., Hogrel, J. Y., & Duchêne, J. (2014). Effect of Different Visual Feedback Conditions on Maximal Grip-Strength Assessment. In XIII Mediterranean Conference on Medical and Biological Engineering and Computing 2013 (pp. 1127-1131). Springer, Cham.